CLINICAL TRIAL: NCT04576364
Title: 12-hour Versus 24-hour Postpartum Magnesium Sulphate for Preeclamptic Patients :A Randomized Controlled Trial
Brief Title: 12-hour Versus 24-hour Postpartum Magnesium Sulphate for Preeclamptic Patients
Acronym: Mgso4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mai Mahmoud Mohamed, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Postpartum Mgso4
Record Dates: First submitted 2020-09-28; First posted 2020-10-06 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Maternal Care Patterns
MeSH Terms: interventions — Magnesium Sulfate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 12-hour postpartum Mgso4 (Active Comparator): Patients having preeclampsia with severe features will receive 12-hour postpartum Mgso4
  Interventions: Drug: Magnesium sulfate for 12 hour
- 24-hour postpartum Mgso4 (Active Comparator): Patients having preeclampsia with severe features will receive 24-hour postpartum Mgso4
  Interventions: Drug: Magnesium sulfate for 24 hour

INTERVENTIONS:
Drug: Magnesium sulfate for 12 hour — drug used to prevent convulsions in patients having preeclampsia with severe features
  Arms: 12-hour postpartum Mgso4
Drug: Magnesium sulfate for 24 hour — drug used to prevent convulsions in patients having preeclampsia with severe features
  Arms: 24-hour postpartum Mgso4

SUMMARY:
To compare the use of magnesium sulfate for 12 hours versus 24 hours in postpartum women with pre-eclampsia with severe features , to ensure maximum efficacy of anticonvulsant action that can be achieved with least exposure to Mgso4 side effects.

DETAILED DESCRIPTION:
Hypertensive disorders of pregnancy constitute one of the leading causes of maternal and perinatal mortality worldwide. It has been estimated that preeclampsia complicates 2-8% of pregnancies globally.

Preeclampsia is a disorder of pregnancy associated with new-onset hypertension, which occurs most often after 20 weeks of gestation and frequently near term. Although often accompanied by new-onset proteinuria, hypertension and other signs or symptoms of preeclampsia may present in some women in the absence of proteinuria. Recently preeclampsia is divided into preeclampsia with severe features, preeclampsia without severe, features. One of serious complication of preeclampsia is occurrence of eclampsia. Eclampsia refers to the occurrence of new-onset, generalized, tonic-clonic seizures or coma in a woman with preeclampsia. Eclampsia can be prevented with magnesium sulphate, which decreases the risk of seizures by 50%, paralleled by a reduction in maternal mortality. It is considered as the gold standard of management of eclampsia Although magnesium sulphate administration is recommended for all women with severe preeclampsia, consensus has not yet to be reached on the ideal duration of prophylactic postpartum anticonvulsant therapy. The use of magnesium sulphate has been recommended for 24 hours following delivery, the period of greatest risk for the occurrence of eclampsia. There are other regimen 12-hour, 6-hour Use of magnesium sulphate therapy is not without complications, consequently longer duration therapy possesses the risk of magnesium toxicity such as respiratory depression, renal and neuromuscular dysfunction. Risks of these complications require regular supervision; hence it is particularly important to assess the minimum effective duration of treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients who have pre-eclampsia with severe features as defined by American College of Obstetricians and Gynecologists guidelines 2019(defined in methodology)
* Singleton pregnancy.
* who accept to participate the study.

Exclusion Criteria:

* Patients with eclampsia
* Epilepsy
* Central Nervous System disorder
* Chronic kidney disease
* Seizures due to metabolic disturbances, space occupying lesions or intra cerebral infections
* Cardiac patients
* Hypersensitivity to Mgso4

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 280 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Need to prolong treatment | up to 12 hour
  Compare efficacy of 12-hour vs 24 hour postpartum Mgso4 in the term of Percentage of patients who will Need to prolong treatment in each group.

SECONDARY OUTCOMES:
Percentage of prevention of eclampsia | up to 24 hour
  Number of patients who develop eclampsia in each group.

CONTACTS AND LOCATIONS:
Overall Officials: ِAhmed Fayek, Proffessor, Study Director — Assiut University; sherif Badran, Lecturer, Study Director — Assiut University
Locations (2):
- Egypt (2):
  - Assuit University women Health hospital, Asyut, Assuit
  - Mai mahoud, Asyut